CLINICAL TRIAL: NCT02009202
Title: Preparation Prior to Colonoscopy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Ewa Idvall, Professor, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS60-12/567
Record Dates: First submitted 2013-11-28; First posted 2013-12-11 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Colon preparation; Child
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Polyethylene Glycols; picosulfate sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- picosulphate (Active Comparator): Picosulphate is given orally
  Interventions: Drug: picosulphate
- polyethylene glycol (Active Comparator): Polyethylene glycol is given orally
  Interventions: Drug: polyethylene glycol

INTERVENTIONS:
Drug: polyethylene glycol
  Arms: polyethylene glycol
Drug: picosulphate
  Arms: picosulphate

SUMMARY:
Colonoscopy is a routinely performed examination of children and adolescents in the diagnostic process of inflammatory bowel disease (IBD). It is necessary that the bowel is clean so the colonoscopy can be optimally performed. The cleansing of the bowel by means of laxatives prior to the examination is, however, considered difficult by many children. Getting smaller children to cooperate and to drink a substantial volume of laxative fluid prior to the examination can be particularly difficult. There are several possible cleansing procedures and combinations of procedures for the cleansing of the colon, for example by means of polyethylene glycol and sodium picosulphate, which are the two most commonly used methods. Cleansing by means of polyethylene glycol can, due to the necessary intake of a substantial quantity of fluid, be particularly frustrating for patients. Often the only way to carry out the preparation is with the insertion of a nasogastric tube, which can cause discomfort for some children. Cleansing the colon by means of sodium picosulphate, which involves an intake of a small quantity of fluid, has been suggested to be a good sufficient method resulting with a satisfactory result in terms of bowel cleanliness. However, studies have so far encompassed only a smaller number of children and further studies are needed to confirm that there is no difference between the two methods in terms of resultant bowel cleanliness.

The purpose of this randomized controlled study is to compare preparation by means of polyethylene glycol and preparation with sodium picosulphate prior to colonoscopy in children.

One hundred children scheduled for colonoscopy in southern Sweden will be randomized into either patient group 1 (for preparation with polyethylene glycol) or patient group 2 (for preparation with sodium picosulphate). For the random sampling, data-driven selection will be implemented. A CONSORT Flowchart (2012) will be encompassed by the study. To assess the cleanliness of the intestinal tract (and volume of fluid in the intestine), the Ottawa Scale will be used (Rostom & Jolicoeur, 2009). All colonoscopy examinations will be performed by the same paediatric gastroenterologist, to whom no information about which preparation method was used by each child will be disclosed. Furthermore, the gastroenterologist will, meet with the children first after the investigation has been completed. All information regarding the investigation will be given to the patient by the admitting physician. During the colonoscopy the gastroenterologist will evaluate the intestinal cleanliness and submit the reports in sealed coded envelopes to the nurse in charge of the patient.

ELIGIBILITY:
Inclusion Criteria:

* elective colonoscopy

Exclusion Criteria:

* not Swedish speaking

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clean colon/Ottowa scale | The day of colonoscopy.
  "Clean colon" will be assessed when the colonoscopy is done.

SECONDARY OUTCOMES:
Patient reported outcome measures | The day of colonoscopy and after 1 week
  Patient questionnaire: 11 questions to be answered by the patients x 2. And further 2 questions the day of colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Idvall, Professor, Principal Investigator — Malmö University
Locations (1):
- Malmö University, Malmo, Skåne County, Sweden

REFERENCES:
- [Derived] Vejzovic V, Wennick A, Idvall E, Agardh D, Bramhagen AC. Polyethylene Glycol- or Sodium Picosulphate-Based Laxatives Before Colonoscopy in Children. J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):414-9. doi: 10.1097/MPG.0000000000000978. PMID 26360658